CLINICAL TRIAL: NCT00379626
Title: Cognitive Group and Hormonal Treatment of Sex Offenders.
Brief Title: Cognitive and Hormonal Treatment of Sex Offenders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: too few patients participated
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH 048-01
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Paraphilia
Keywords: Paraphilia; Hormonal treatment; Cognitive treatment
MeSH Terms: conditions — Paraphilic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive and hormone treatment (Experimental): cognitive and hormone (Leuprorelin) treatment
  Interventions: Drug: cognitive and hormone treatment

INTERVENTIONS:
Drug: cognitive and hormone treatment — cognitive and hormone (Leuprorelin) treatment

SUMMARY:
The aim of this study is to determine if Cognitive treatment and hormone treatment can change the relapse rate of sexual offenders.

DETAILED DESCRIPTION:
The aim of this study is to determine if Cognitive treatment and hormone treatment can change the relapse rate of sexual offenders.

In the first part of study we are studying changes in the offenders cognitive distortions and in the second part we are studying changes in sexual activities and sexual thoughts after treatment with Leuprorelin. The study is an open pre and post study.

ELIGIBILITY:
Inclusion Criteria:

Men sentenced for paraphilia

Exclusion Criteria:

Men above 70 years and men that does not speak english

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The degree of cognitive distortions after treatment | 8 months

SECONDARY OUTCOMES:
Locus of control after treatment in part one. | 8 months
Degree of mental health problems (SCL-90) | 8 months
The testosterone levels before, during and after treatment | baseline upto 8 months
  measured each 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Jim Aa Nøttestad, Dr. Philos, Principal Investigator — St. Olavs Hospital, Departement of forensic psychiatry, Brøset
Locations (1):
- St. Olavs Hospital. Departement for forensic psyciatry, Brøset., Trondheim, Norway

REFERENCES:
- [Result] Nottestad JA, Bjarnar E, Lundmo PI, Sandvik M. [Treatment of sex offenders with leuprorelin]. Tidsskr Nor Laegeforen. 2006 Feb 23;126(5):633-4. No abstract available. Norwegian. PMID 16505878